CLINICAL TRIAL: NCT05366621
Title: The Association Between Anti-osteoporosis Medications and Lowered All Cause Mortality After Osteoporotic Fractures
Brief Title: Post-fracture Medication and Mortality
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Hsing Wu, Associate Professor, National Cheng-Kung University Hospital
Other Study IDs: Osteoporosis and Mortality
Record Dates: First submitted 2022-05-02; First posted 2022-05-09 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Osteoporosis; Osteoporosis Fracture; Drug Therapy; Mortality; Adherence, Medication
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures; Medication Adherence | interventions — Diphosphonates; Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Used osteoporosis medication: Patients who had used osteoporosis medication after osteoporotic fractures.
  Interventions: Drug: Anti-osteoporosis medications
- Did not use osteoporosis medication: Patients who didn't use osteoporosis medication after osteoporotic fractures.
  Interventions: Drug: Anti-osteoporosis medications

INTERVENTIONS:
Drug: Anti-osteoporosis medications — Medication exposure was defined as the usage of osteoporosis medications approved by the Taiwan Food and Drug Administration (TFDA), including alendronate, risedronate, ibandronate, zoledronic acid, denosumab, raloxifene, bazedoxifene, calcitonin, and teriparatide, but excluded patients using the osteoporosis medication for cancer-related treatments (such as high dosing frequency of zoledronic acid or denosumab).
  Other Names: Bisphosphonates; Denosumab; Hormone-related therapy; Bone-building medication

SUMMARY:
Osteoporotic fracture is a common public-health problem in the whole world. Although postfracture usage of anti-osteoporosis medications, may reduce mortality, recent results have been inconsistent. The investigators aim to examine associations between osteoporosis medication and mortality in older adults and any type of fracture patients. The investigators also aim to discuss the pleiotropic effects of different types of anti-osteoporosis medications.

DETAILED DESCRIPTION:
Osteoporotic fracture has become a serious health and economic burden as life expectancy increases. In a WHO report, the burden of osteoporotic fractures in 2002 was 2.8 million disability-adjusted life years, which is more than that for hypertension and slightly less than that for diabetes mellitus or chronic obstructive pulmonary diseases. Many patients who have had a diagnosed fracture have never been diagnosed with osteoporosis, therefore, closing the gap in osteoporosis treatment is important. This situation is primarily due to the fact that osteoporosis symptoms are often not recognized until a fracture occurs. Osteoporotic fractures, especially those of the hip and vertebral, are associated with an increased risk of death. Early detection of high risk for osteoporotic fractures is important; however, post-fracture management, especially interventions intended to lower mortality, is an emerging public health issue in rapidly aging societies. The burden of osteoporotic fracture is higher than that of hypertension, however, osteoporosis is always given less attention than other chronic diseases by health professionals and the general population.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed osteoporosis and hip fracture are defined as a claim record from the NHIRD between 2009 and 2017.

Exclusion Criteria:

* Patients with a diagnosis of osteoporosis or osteoporotic fractures in 2008 or before were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The final study participants included those who satisfied the inclusion criteria for both osteoporosis and hip fracture cohorts, and they were followed until 2018.
Sampling Method: Non-Probability Sample
Enrollment: 216155 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of deaths with and without anti-osteoporotic therapy after hip fracture surgery | 12 years
  This is the number of participants who died during the time of observation from Taiwan's National Health Insurance Research Database.
Number of deaths with or without anti-osteoporosis therapy after hip or vertebral fracture surgery among older adults | 12 years
  This is the number of participants who died during the time of observation from Taiwan's National Health Insurance Research Database.
Number of deaths with and without bisphosphonates after hip or spine fracture surgery | 12 years
  This is the number of participants who died during the time of observation from Taiwan's National Health Insurance Research Database.
Number of deaths with different types of anti-osteoporosis treatments after post-fracture | 12 years
  This is the number of participants who died during the time of observation from Taiwan's National Health Insurance Research Database.
Number of deaths in five leading causes of death with and without anti-osteoporosis treatment after post-fracture | 12 years
  This is the number of participants who died during the time of observation from Taiwan's National Death Registry. The five leading causes are defined as the main five leading causes.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsing Wu, MD, Study Director — National Cheng Kung University
Locations (1):
- Department of Family Medicine, National Cheng Kung Univ Hosp, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No